CLINICAL TRIAL: NCT00556140
Title: The Combination of Aripiprazole and Selective Serotonin Reuptake Inhibitor (SSRI) Antidepressants in the Acute Treatment of Psychotic Major Depression: Efficacy and Tolerability
Brief Title: The Combination of Aripiprazole and Antidepressants in Psychotic Major Depression
Acronym: Abilify
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, John D. Matthews, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003-P-000990
Record Dates: First submitted 2007-11-08; First posted 2007-11-09 (Estimated); Results first posted 2012-08-20 (Estimated); Last update posted 2012-08-20 (Estimated); Status verified 2012-07

CONDITIONS: Psychotic Depression
MeSH Terms: interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Major Depression with Psychotic Features (Experimental)
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole — Everyone in this study will receive aripiprazole and an antidepressant called a selective serotonin reuptake inhibitor (SSRI). There is only one arm for this study.
  Aripiprazole is an antipsychotic medication that has been approved by the Food and Drug Administration (FDA) for the treatment of schizophrenia.
  You will receive aripiprazole (Abilify) and one of the following SSRI antidepressant medications that will be determined by the study doctor and you: sertraline (Zoloft), citalapram (Celexa), or escitalopram (Lexapro). The dose of aripiprazole (Abilify) will be 10 milligrams a day, and the starting doses for the SSRI anti-depressants will be: sertraline (Zoloft) 50 milligrams a day, citalopram (Celexa) 20 milligrams a day, and escitalopram (Lexapro) 10 milligrams a day.
  Other Names: Abilify

SUMMARY:
The purpose of the study is to assess the safety and effectiveness of the combination of aripiprazole (Abilify) and selective serotonin reuptake inhibitors (SSRIs) in subjects with psychotic major depression.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18-80 years, inclusive.
2. Drug-free outpatients or inpatients meeting DSM-IV criteria for major depression with psychotic features.
3. Inpatients who undergo a 5-7 day washout period of their medication while concurrently beginning one of the approved SSRI's and abilify.
4. HAM-D-24 score > 16.

Exclusion Criteria:

1. Pregnant women and women of child bearing potential not using a medically accepted means of contraception (oral contraceptives are allowed).
2. Women who are breast-feeding.
3. Patients meeting DSM-IV criteria for major depression without psychotic features, or psychosis without major depression at the screen visit.
4. Patients with serious suicidal risk.
5. Patients with a history of seizure disorder; unstable physical disorders (cardiovascular, hepatic, renal, respiratory, endocrine, neurologic, or hematologic); or any physical disorder judged to significantly affect central nervous system function.
6. Patients meeting criteria for the following DSM-IV diagnoses: organic mental disorders; substance use disorders, including alcohol, active within the last 6 months; bipolar disorder; schizoaffective disorder; or antisocial personality disorder.
7. Patients who are currently taking an antidepressant, antipsychotic, or mood stabilizing drug and who are responding to one or all of these medications. If patients are not responding to these medications, they may go through a washout period of at least one week under the supervision of a study doctor before entering into this study.
8. Patients who are not able to read and understand the consent form, or who are not capable of understanding or giving informed consent to the procedures of the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2003-06; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthews D John, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Matthews JD, Siefert C, Dording C, Denninger JW, Park L, van Nieuwenhuizen AO, Sklarsky K, Hilliker S, Homberger C, Rooney K, Fava M. An open study of aripiprazole and escitalopram for psychotic major depressive disorder. J Clin Psychopharmacol. 2009 Feb;29(1):73-6. doi: 10.1097/JCP.0b013e318193dfb4. PMID 19142112

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment ran from Sept. 13, 2004 to Aug. 9, 2006 from the Massachusetts General Psychiatry Inpatient and Outpatient clinics.
Pre-assignment Details: All participants enrolled in the study were given aripiprazole and escitalopram.
Groups:
- Major Depression With Psychotic Features: All patients received aripiprazole 10 milligrams and escitalopram 10 milligrams as starting doses. These doses were increased to 20 milligrams and 30 milligrams, respectively. These increases occurred over a period of 7 weeks.
Period: Overall Study
Arm/Group | Major Depression With Psychotic Features
Started | 16
Completed | 13
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Major Depression With Psychotic Features
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 41.8 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Depression and Psychosis Response Rate
Description: This response rate refers to the percentage of patients who experienced a 50 percent or greater reduction in symptoms. Specifically, this refers to a 50 percent reduction in Hamilton Depression Rating Scale 17 (HAM-D-17) scores from baseline and no psychotic symptoms as measured by the Structured Clinical Interview for DMS-IV psychosis module. HAM-D-17 scores range from 0-50 with a score of >23 considered severely depressed and <7 to be mildly to not at all depressed.
Time Frame: Baseline and 7 weeks
Population: For the 3 participants who did not complete the study, the "last observation carried forward" technique was used to replace missing data for them.
Measure: Number; unit: percent of participants
Arm/Group | Major Depression With Psychotic Features
Number analyzed (Participants) | 16
percent of participants | 62.5 (8.3)

2. Secondary Outcome: Depression and Psychosis Remission Rate
Description: This remission rate refers to a Hamilton Depression Rating Scale 17 (HAM-D-17) score of 7 or less and no psychotic symptoms as measured by the Structured Clinical Interview for DMS-IV psychosis module. HAM-D-17 scores range from 0-50 with a score of >23 considered severely depressed and <7 to be mildly to not at all depressed.
Time Frame: Baseline and 7 weeks
Population: as for outcome 1
Measure: Number; unit: percent of participants
Arm/Group | Major Depression With Psychotic Features
Number analyzed (Participants) | 16
percent of participants | 50

ADVERSE EVENTS:
Arm/Group | Major Depression With Psychotic Features
Serious Adverse Events (participants affected / at risk) | 2/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Major Depression With Psychotic Features (N=16)
Orthostatic hypotension (Vascular disorders) | 1 (1) — 1 subject had a severe orthostatic drop in her blood pressure requiring an ED visit while on aripiprazole 15mg a day, escitalopram 10 mg a day, and propanolol 10 mg 3 times a day.
worsening of major depression with psychotic features (Psychiatric disorders) | 1 (1) — 1 subject had to be hospitalized for worsening of major depression with psychotic features.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Major Depression With Psychotic Features (N=16)
Akathisia (Nervous system disorders) | 10 (10)
Gastrointestinal distress (Gastrointestinal disorders) | 4 (4)
Fatigue (General disorders) | 2 (2)
Sedation (General disorders) | 2 (2)
Body aches (General disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
We had several limitations to the study. The sample size was small, and we used an open and uncontrolled study design. We also excluded subjects who currently or recently abused alcohol, recreational drugs, and/or prescription drugs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes